CLINICAL TRIAL: NCT03090282
Title: Subgingival Microbiome Following Mechanical Treatment and it's Effect on Peri-implant Sub-mucosa in Aggressive Periodontitis Patients
Brief Title: Subgingival Microbiota Following Mechanical Treatment and it's Effect on Peri-implant Sub-mucosa in Periodontitis Patients
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Liu guojing, Principal Investigator, Peking University
Other Study IDs: PKUSSIRB-201525102
Record Dates: First submitted 2017-03-09; First posted 2017-03-24 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Aggressive Periodontitis, Generalized
Keywords: mechanical treatment; implant
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Root Planing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — some bacteria DNA from subgingival. No need for human DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: mechanical treatment(mainly scaling and root planing), periodontal surgery(if indicated), implant placement. — The investigators shall follow the regular procedure to these patients.

SUMMARY:
The investigators planed to observe the microbiome of an aggressive periodontitis patient, during mechanical treatment, surgery(if indicated) and implant placement. The investigators designed to observe the changes after mechanical treatment.Then, the investigators will compare the sub-mucosa microbiome of implant and the subgingival community. The investigators expected a different community after treatment, and there could be similarity between implant and nature teeth.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects were between 18-35 years old and diagnosed with generalized aggressive periodontitis (GAgP) according to the 1999 International Classification of Periodontal Diseases (Armitage 1999);
2. At least 20 teeth in the first appointment and at least 3 teeth(other than first molars and central incisors)with a probing depth(PD) ≥ 6mm, clinical attachment level (CAL)≥5mm;
3. The clinical diagnosis was confirmed by evidence of inter-proximal bone loss on full-mouth periapical radiographs;
4. Family history of aggressive periodontitis.

Exclusion Criteria:

1. Uncontrolled systemic conditions including diabetes and hypertension;
2. Pregnant or lactating;
3. Smoking;
4. Received periodontal treatment within the previous 6 months or antibiotic medication during the previous 3 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: aggressive periodontitis patients with defection of dentition or shall extracted hopeless teeth, and intended to implant treatment.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
changes of diversity of subgingival community (compare the sub-mucosa microbiome of implant and the subgingival community) | Baseline, 6 weeks after mechanical treatment
  the diversity of subgingival community before and after mechanical treatment
changes of diversity of subgingival community (compare the sub-mucosa microbiome of implant and the subgingival community) | before implantation, 1 months after second stage surgery, and every month after prosthetic treatment until 2 years.
  the diversity of submucosa community before and after implatation
changes of prevalence and abundance of OTUs | Baseline, 6 weeks after mechanical treatment
  compute and compare the prevalence and abundance of OTUs
changes of prevalence and abundance of OTUs | before implantation, 1 months after second stage surgery, and every month after prosthetic treatment until 2 years.
  compute and compare the prevalence and abundance of OTUs

SECONDARY OUTCOMES:
changes of bleeding index | Baseline, 6 weeks after mechanical treatment, before implantation, 1 months after second stage surgery, every month after prosthetic treatment until 2 years.
  bleeding index after probing
changes of probing depth | Baseline, 6 weeks after mechanical treatment, before implantation, 1 months after second stage surgery, every month after prosthetic treatment until 2 years.
  probing depth of indicated sites
clinical attachment loss | Baseline, 6 weeks after mechanical treatment, before implantation, 1 months after second stage surgery, every month after prosthetic treatment until 2 years.
  by probe, the distance between CEJ and gingival sulcus

CONTACTS AND LOCATIONS:
Overall Officials: Yu xiaoqian, Study Chair — Peking University Hospital of Stomatology; Liu guojing, Principal Investigator — Peking University Hospital of Stomatology
Locations (1):
- Peking university hospital of stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
haven't decided yet

REFERENCES:
- [Derived] Liu G, Luan Q, Chen F, Chen Z, Zhang Q, Yu X. Shift in the subgingival microbiome following scaling and root planing in generalized aggressive periodontitis. J Clin Periodontol. 2018 Apr;45(4):440-452. doi: 10.1111/jcpe.12862. Epub 2018 Mar 6. PMID 29266363